CLINICAL TRIAL: NCT00945724
Title: A Phase II Study of R-CHOP With Intensive CNS Prophylaxis and Scrotal Irradiation in Patients With Primary Testicular Diffuse Large B-cell Lymphoma
Brief Title: Safety and Feasibility Study of Combination of State of Art Chemoimmunotherapy, Intensive Central Nervous System Prophylaxis and Scrotal Irradiation to Treat Primary Diffuse Large B-cell Lymphoma of Testis
Acronym: IELSG30
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG30; EudraCT Number 2009-011789-26
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Large B-cell Diffuse Lymphoma of Testis
MeSH Terms: interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; Methotrexate

ARMS (1):
- R-CHOP, Depocyte, Methotrexate (Experimental)
  Interventions: Drug: Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisolone, liposomal cytarabine, methotrexate

INTERVENTIONS:
Drug: Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisolone, liposomal cytarabine, methotrexate — Weeks 1-15:
  * 6 cycles of CHOP on Days 1 to 5, to be repeated q21 Days
  * Rituximab 375 mg/m2 on Day 0 or Day 1 of every CHOP cycle
  * IT chemoth:Depocyte 50 mg on Day 0 of cycles 2,3,4&5 of R-CHOP
  Weeks 18-22:
  • Methotrexate 1.5 g/m2 q14 Days x 2
  From Week 24:
  • Scrotal prophylactic radiotherapy or involved field radiotherapy(but can be planned concomitantly to R-CHOP in pts with bilateral disease)

SUMMARY:
This trial is a phase II non-comparative study aimed to determine the feasibility and toxicity of the R-CHOP regimen in combination with intrathecal liposomal cytarabine and systemic intermediate-dose methotrexate followed by loco-regional radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary testicular lymphoma at diagnosis. Histological subtype included into the study is only Diffuse Large B Cell Lymphoma (Attachment 2: WHO classification of lymphoma).
2. Orchiectomy is mandatory, before enrolment of the patient into the study.
3. Orchiectomy should be performed within 2 months before study entry.
4. Age 18-80
5. Untreated patients
6. Ann Arbor Stage IE and IIE. Bilateral testicular involvement at presentation will not be considered Stage IV. These patients may be included into the study and the final Ann Arbor stage (I or II) will be determined by the extent of nodal disease.
7. Bidimensionally measurable or evaluable disease. Patients who have had all disease removed by surgery are eligible.
8. Adequate haematological counts: ANC > 1.0 x 109/L and PLTs count > 75 x 109/L
9. Cardiac ejection fraction ≥ 45% by MUGA scan or echocardiography
10. Non peripheral neuropathy or any active non-neoplastic CNS disease.
11. No other major life-threatening illnesses that may preclude chemotherapy
12. Conjugated bilirubin ≤ 2 x ULN.
13. Alkaline phosphatase and transaminases ≤ 2 x ULN.
14. Creatinine clearances ≥ 45 ml/min.
15. HIV negativity
16. HBV negativity or patients with HBVcAb +, HbsAg -, HBs Ab+/- with HBV-DNA negative
17. HCV negativity with the exception of patients with no signs of active chronic hepatitis histologically confirmed
18. Life expectancy > 6 months.
19. Performance status < 2 according to ECOG scale.
20. No psychiatric illness that precludes understanding concepts of the trial or signing informed consent
21. Written informed Consent

Exclusion Criteria:

1. Has known or suspected hypersensitivity or intolerance to rituximab
2. History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
3. Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug)
4. Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 5, NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
5. History of clinically relevant hypotension
6. CNS involvement (meningeal and/or brain involvement by lymphoma)
7. Evolving malignancy within 3 years with the exception of localized non-melanomatous skin cancer
8. HIV positivity
9. HBV positivity with the exception of patients with HBVcAb +, HbsAg -, HBs Ab+/- with HBV-DNA negative
10. HCV positivity with the exception of patients with no signs of active chronic hepatitis histologically confirmed
11. Active opportunistic infection
12. Receipt of extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy
13. Exposure to Rituximab prior study entry
14. Have received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study.
15. Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-09-27 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Zucca, MD, Study Chair — IOSI
Locations (22):
- Italy (21):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Spedali Civili, Brescia
  - Ematologia Ospedale Businco, Cagliari
  - S. Martino Hospital, Genova
  - European Institute of Oncology, Milan
  - San Raffaele H Scientific Institute, Milan
  - Policlinico, Modena
  - A.O. San Gerardo, Monza
  - AOU Maggiore della Carità, Novara
  - S. Matteo, Pavia
  - Ospedale Civile, Piacenza
  - U.O. Ematologia AUSL Ravenna, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - IFO Regina Elena, Roma
  - Policlinico Universitario Campus Biomedico, Roma
  - Università La Sapienza, Rome
  - Humanitas, Rozzano
  - Azienda Ospedaliero-Universitaria, Sassari
  - A.O. S. Maria, Terni
  - A.O.U. San Giovanni Battista-Molinette, S.C. Ematologia 2, Torino
  - Ospedale di Circolo Fondazione Macchi, Varese
- IOSI, Bellinzona, Switzerland

REFERENCES:
- [Derived] Conconi A, Chiappella A, Ferreri AJM, Stathis A, Botto B, Sassone M, Gaidano G, Balzarotti M, Merli F, Tucci A, Vanazzi A, Tani M, Bruna R, Orsucci L, Cabras MG, Celli M, Annibali O, Liberati AM, Zanni M, Ghiggi C, Pisani F, Pinotti G, Dore F, Esposito F, Pirosa MC, Cesaretti M, Bonomini L, Vitolo U, Zucca E. IELSG30 phase 2 trial: intravenous and intrathecal CNS prophylaxis in primary testicular diffuse large B-cell lymphoma. Blood Adv. 2024 Mar 26;8(6):1541-1549. doi: 10.1182/bloodadvances.2023011251. PMID 38181782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment lasted from 27 September 2009 to 13 July 2017
Period: Overall Study
Arm/Group | R-CHOP, Depocyte, Methotrexate
Started | 54
Completed | 45
Not Completed | 9
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Adverse Event | 5
Not completed — Second malignancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | R-CHOP, Depocyte, Methotrexate
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 27
Age, Continuous [Median (Full Range); unit: years] | 66 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 47
  Switzerland | 7
Ann Arbor stage [Count of Participants; unit: Participants] — Ann Arbor staging is the staging system for lymphomas. The stage depends on the place where the malignant tissue is located.
  * Stage I indicates that the cancer is located in a single region, usually one lymph node and the surrounding area.
  * Stage II indicates that the cancer is located in two separate regions, an affected lymph node or lymphatic organ and a second affected area, both affected areas are confined to one side of the diaphragm.
  Stage II indicates a worse outcome.
  Participants
    Stage I | 32
    Stage II | 22
Bilateral testicular location [Count of Participants; unit: Participants]
  Bilateral testicular location | 1
  No bilateral testicular location | 53
B symptoms [Count of Participants; unit: Participants] — B symptoms include fever, night sweats and weight loss of ≥10% of body weight over 6 months. Presence of B symptoms indicates a worse outcome.
  Participants
    Presence of B symptoms | 2
    No Presence of B symptoms | 52
Serum lactate dehydrogenase (LDH) [Count of Participants; unit: Participants]
  > normal upper value | 7
  </= normal upper value | 47
Serum Beta2-microglobulin [Count of Participants; unit: Participants]
  > normal upper value | 8
  </= normal upper value | 40
  Not recorded | 6

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Assessment
Description: Number of patients who withdrew the treatment due to adverse event
Time Frame: From treatment start until the last drug administration, up to week 22 for the 'R-CHOP, Depocyte, Methotrexate' Group, up to 15 weeks (Weeks 1-15) for the 'R-CHOP + Lyposomal Cytarabine' Group, and from week 18-22 for the 'HD-MTX' Group
Population: Weeks 1 -15 All patients treated with 6 cycles of R-CHOP (CHOP21) on days 0/1 to 5, to be repeated every 21 days Intratecal (IT) Chemotherapy: liposomal cytarabine on day 0 of cycles 2, 3, 4 and 5 of R-CHOP Weeks 18 - 22 High Dose (HD) Methotrexate (MTX) Days 0 - 4 of two 14 days cycles From Week 25 Scrotal prophylactic radio therapy (RT) to the contralateral testis.
Measure: Count of Participants; unit: Participants
Groups:
- R-CHOP + Lyposomal Cytarabine: Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisolone, liposomal cytarabine, methotrexate: Weeks 1-15:
  * 6 cycles of CHOP on Days 1 to 5, to be repeated q21 Days
  * Rituximab 375 mg/m2 on Day 0 or Day 1 of every CHOP cycle
  * IT chemoth:Depocyte 50 mg on Day 0 of cycles 2,3,4&5 of R-CHOP
- HD-MTX: Weeks 18-22:
  • Methotrexate 1.5 g/m2 q14 Days x 2
Arm/Group | R-CHOP, Depocyte, Methotrexate | R-CHOP + Lyposomal Cytarabine | HD-MTX
Number analyzed (Participants) | 54 | 54 | 48
Participants | 6 | 3 | 3

2. Secondary Outcome: 5 Year Cumulative Incidence of Progressions
Description: Percentage of patients with disease progression after achieving a remission
Time Frame: From the first documented response to relapse until 5 years from study entry
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP, Depocyte, Methotrexate
Number analyzed (Participants) | 54
percentage of participants | 6 [2 to 16]

3. Secondary Outcome: 5 Years Progression Free Survival (PFS)
Description: Percentage of patients free from disease progression after 5 years from study entry
Time Frame: From study entry until 5 years after
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP, Depocyte, Methotrexate
Number analyzed (Participants) | 54
percentage of participants | 91 [79 to 96]

4. Secondary Outcome: 5 Years Overall Survival (OS)
Description: Percentage of patients alive after 5 years from study entry
Time Frame: From study entry until 5 years after
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP, Depocyte, Methotrexate
Number analyzed (Participants) | 54
percentage of participants | 92 [81 to 97]

ADVERSE EVENTS:
Time Frame: All cause mortality was assessed through 5 years after study entry. All AEs were collected from the date of informed consent signature until 30 days after the end of treatment (week 26) for the "R-CHOP, Depocyte, Methotrexate" group; from the date of informed consent signature up to week 17 for the 'R-CHOP + Lyposomal Cytarabine' Group; from week 18 until 30 days after the end of treatment (week 26) for the 'HD-MTX' Group
Description: SAE suspected to be related to the study treatment that occurred after the defined reporting period and up to 8 years from treatment start had also to be reported to the Sponsor.
Groups:
- Safety Population: All patients who have received at least one dose of treatment will be considered as Safety Population
- R-CHOP + Lyposomal Cytarabine: Subjects treated with R-CHOP (CHOP21).
- HD-MTX: Subjects treated with HD-MTX.
Arm/Group | Safety Population | R-CHOP + Lyposomal Cytarabine | HD-MTX
All-Cause Mortality (participants affected / at risk) | 12/54 | 0/54 | 0/48
Serious Adverse Events (participants affected / at risk) | 19/54 | 17/54 | 3/48
Other Adverse Events (participants affected / at risk) | 47/54 | 47/54 | 17/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=54) | R-CHOP + Lyposomal Cytarabine (N=54) | HD-MTX (N=48)
Increase of neutrophilis (Investigations) | 1 (1) | 1 (1) | 0 (0)
Prostatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac general pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 0 (0)
Mucositis (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction/extravasation changes (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Acute urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=54) | R-CHOP + Lyposomal Cytarabine (N=54) | HD-MTX (N=48)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 7 (13) | 8 (10) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 12 (19) | 11 (15) | 2 (3)
Diarreha (Gastrointestinal disorders) | 7 (11) | 6 (9) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (3) | 0 (0)
Fatigue (General disorders) | 9 (20) | 8 (16) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 0 (0)
Fever (General disorders) | 11 (17) | 9 (14) | 3 (3)
Flue-like Syndrome (General disorders) | 4 (4) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 14 (20) | 14 (19) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 7 (21) | 6 (17) | 3 (3)
Mucositis (General disorders) | 6 (7) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 9 (20) | 9 (17) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 21 (34) | 17 (28) | 4 (4)
Pain (General disorders) | 10 (16) | 10 (12) | 2 (3)
Paresthesia (Nervous system disorders) | 6 (7) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Sensitive/Peripheral Neuropathy (Nervous system disorders) | 7 (7) | 6 (6) | 1 (1)
Transaminases increase (Hepatobiliary disorders) | 7 (12) | 6 (10) | 2 (2)
Trombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-05-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT00945724/Prot_SAP_000.pdf